CLINICAL TRIAL: NCT00585416
Title: A Phase II Study of CGC-11047 in Patients With Metastatic Hormone Refractory Prostate Cancer (47-02-001)
Brief Title: Study of CGC-11047 in Patients With Metastatic Hormone Refractory Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Further evaluation of phase I dosing
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Progen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC2006-0099; CO06801; 47-02-001
Record Dates: First submitted 2007-12-21; First posted 2008-01-03 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2009-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Hormone Refractory; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — CGC 11047

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): CGC-11047 IV weekly for 3 weeks followed by one rest week (4weeks=1cycle)
  Interventions: Drug: CGC-11047

INTERVENTIONS:
Drug: CGC-11047 — CGC-11047 IV weekly for 3 weeks followed by one rest week (4weeks=1cycle)

SUMMARY:
The purpose of this research is to determine the effectiveness of CGC-11047 in subjects with metastatic hormone refractory prostate cancer as measured by changes in PSA.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic hormone refractory prostate cancer.
* Eastern Cooperative Oncology Group (ECOG) Performance status of 0-1.
* testosterone <50ng/dL. Patients must continue primary androgen deprivation with an LHRH analogue if they have not undergone orchiectomy.
* Progressive disease after androgen deprivation.

Exclusion Criteria:

* Patients whose clinical condition would make chemotherapy clearly indicated.
* Patients who have received systemic chemotherapy for the treatment of metastatic disease.
* Peripheral neuropathy > Grade 1
* Prior anti-angiogenic therapy, including thalidomide.
* Patients with inadequate recovery from any prior surgical procedure, or patients having undergone any major surgical procedure or radiation within 4 weeks prior to study entry.
* Patients who have received radiopharmaceuticals (strontium, samarium) within 8 weeks prior to enrollment.
* Patients with known brain metastases or history of brain metastases.
* History of stroke within 6 months of treatment or other significant neurological limitations.
* Patients who have received more than 2 prior investigational treatments.
* Uncontrolled intercurrent illness
* Patients with a history of a myocardial infarction within the prior 6 months or, hospitalizations for decompensated congestive heart failure within the prior 6 months, or history of significant / symptomatic cardiac arrhythmias

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Efficacy | 8 weeks

SECONDARY OUTCOMES:
Safety | Throughout and for 28 days post drug

CONTACTS AND LOCATIONS:
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States